CLINICAL TRIAL: NCT02687035
Title: The PARTNER II Trial: Placement of AoRTic TraNscathetER Valves: Continued Access Program for SAPIEN 3 Intermediate Risk (S3iCAP)
Brief Title: PARTNER II Trial: S3iCAP
Acronym: PII S3i CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-12 S3iCAP
Record Dates: First submitted 2016-02-01; First posted 2016-02-22 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-12

CONDITIONS: Aortic Stenosis
Keywords: S3iCAP; SAPIEN 3; Transfemoral; Commander; Certitude; TAVR; TAVI; Aortic stenosis; THV; Transcatheter Heart Valve; TVT; TVTR
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TAVR (Experimental): Intermediate risk patients receiving transcatheter aortic valve replacement (TAVR)
  Interventions: Device: SAPIEN S3 valve

INTERVENTIONS:
Device: SAPIEN S3 valve — Transcatheter aortic valve replacement
  Other Names: TAVR; TAVI; Transcatheter aortic valve replacement; SAPIEN

SUMMARY:
Following completion of enrollment in the PARTNER II SAPIEN 3 intermediate risk trial, this trial provided continued access to treatment for subjects with severe aortic stenosis who were at intermediate surgical risk.

DETAILED DESCRIPTION:
This multi-center, single arm registry will provide continued access of the Edwards SAPIEN 3 Transcatheter Heart Valve and delivery systems to severe aortic stenosis patients at intermediate risk for standard aortic valve replacement. Patient data will be entered into the TVT Registry (TVTR) from screening through 1 year including the collection of 5 year follow-up through CMS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be covered by Medicare. This will enable Edwards to link to the CMS database for long term follow-up through 5 years. No other insurance provider will be accepted.
2. Assessment of intermediate surgical risk defined as STS 4-8% or heart team assessment of intermediate risk factors.
3. Patient has senile degenerative aortic valve stenosis with echocardiographically derived criteria: mean gradient > 40 mmHg or jet velocity greater than 4.0 m/s and an initial aortic valve area (AVA) of < 0.8 cm2 or indexed EOA < 0.5 cm2/m2. Qualifying echo must be within 60 days of the date of the procedure.
4. Aortic valve annulus area range (273mm2-680 mm2) per 3D imaging (echo, CT, or MRI).
5. Patient is symptomatic from his/her aortic valve stenosis, as demonstrated by NYHA Functional Class II or greater.
6. The heart team agrees (and verified in the case review process) that valve implantation will likely benefit the patient.
7. Heart team agrees (a priori) on treatment strategy for concomitant coronary disease (if present).
8. The study patient or the study patient's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
9. The study patient agrees to comply with all required post-procedure follow-up visits including annual visits through 5 years and analysis close date visits, which will be conducted as a phone follow-up.

Exclusion Criteria:

1. Heart team assessment of inoperability (including examining cardiac surgeon).
2. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [(defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)].
3. Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified.
4. Mixed aortic valve disease (aortic stenosis and aortic re-regurgitation with predominant aortic regurgitation >3+).
5. Pre-existing mechanical or bioprosthetic valve in any position.
6. Complex coronary artery disease:

   1. Unprotected left main coronary artery
   2. Syntax score > 32 (in the absence of prior revascularization)
7. Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker or ICD is not considered exclusion criteria.
8. Any patient with a balloon valvuloplasty (BAV) < 30 days of the procedure (unless BAV is a bridge to procedure after a qualifying ECHO).
9. Patients with planned concomitant surgical or transcatheter ablation for atrial fibrillation.
10. Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), thrombocytopenia (Plt < 50,000 cell/mL).
11. Hypertrophic cardiomyopathy with or without obstruction (HOCM).
12. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of screening evaluation.
13. Need for emergency surgery for any reason.
14. Severe ventricular dysfunction with LVEF < 20%.
15. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
16. Active upper GI bleeding within 3 months (90 days) prior to procedure.
17. A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure.
18. Native aortic annulus size < 16 mm or > 28mm as measured by echocardiogram.
19. Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 6 months (180 days) of the procedure.
20. Renal insufficiency (creatinine > 3.0 mg/dL) and/or renal replacement therapy at the time of screening.
21. Estimated life expectancy < 24 months (730 days) due to carcinomas, chronic liver disease, chronic renal dis-ease or chronic end stage pulmonary disease.
22. Expectation that patient will not improve despite treatment of aortic stenosis.
23. Significant aortic disease, including marked tortuosity (hyperacute bend), aortic arch atheroma [especially if thick (> 5 mm), protruding or ulcerated] or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta. (Transfemoral)
24. Iliofemoral vessel characteristics that would preclude safe placement of 14F or 16F introducer sheath such as severe obstructive calcification, severe tortuosity or min-imum average vessel size less than 5.5 mm. (Transfem-oral).
25. Currently participating in an investigational drug or an-other device study. Note: Trials requiring extended fol-low-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
26. Active bacterial endocarditis within 6 months (180 days) of procedure.
27. Evidence of intracardiac mass, thrombus, vegetation, active infection or endocarditis.
28. Inability to tolerate anticoagulation/antiplatelet therapy.
29. For transfemoral approach only: Femoro-iliac vessels < 5.5 mm for the 23 mm and the 26 mm system and < 6.0 mm for the 29 mm system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1822 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susheel Kodali, MD, Principal Investigator — University of Columbia; Vinod Thourani, MD, Principal Investigator — Emory University
Locations (56):
- United States (55):
  - Scripps Green Hospital, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Mercy General Hospital, Sacramento, California
  - University of Colorado Hospital, Denver, Colorado
  - Washington Hospital Center DC, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem Research Institute, Evanston, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Indiana University Health-Methodist Hospital, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc./ St. Vincent Heart Center of Indiana, LLC, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville Jewish Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic-Saint Marys Hospital, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City Mid America, Kansas City, Missouri
  - Washington University/ Barnes-Jewish Hospital, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop-University Hospital, Mineola, New York
  - Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Northshore Long Island Jewish Health System, New York, New York
  - Medical University of South Carolina Charleston, Charleston, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Providence Heart & Vascular Institute, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Austin Heart, PLLC, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- St. Paul's Hospital, Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbas AE, Ternacle J, Pibarot P, Xu K, Alu M, Rogers E, Hahn RT, Leon M, Thourani VH. Impact of Flow on Prosthesis-Patient Mismatch Following Transcatheter and Surgical Aortic Valve Replacement. Circ Cardiovasc Imaging. 2021 Aug;14(8):e012364. doi: 10.1161/CIRCIMAGING.120.012364. Epub 2021 Aug 13. PMID 34387097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from January 2015 to August 2016. Subjects in this trial were entered into the TVT Registry. Of the 1822 subjects enrolled in the trial, 1814 subjects received the study device.
Pre-assignment Details: Participants that did not receive an Edwards device were not followed in the trial.
Groups:
- SAPIEN 3: Patients at intermediate surgical risk receiving the SAPIEN S3 valve with Commander or Certitude delivery system.
Period: Overall Study
Arm/Group | SAPIEN 3
Started | 1822
Completed | 1638
Not Completed | 184
Not completed — Withdrawal by Subject | 1
Not completed — Death | 87
Not completed — Lost to Follow-up | 1
Not completed — Missed Visit | 87
Not completed — Did not receive Study Device | 8

BASELINE CHARACTERISTICS:
Population: 1814 subjects received the SAPIEN 3 valve
Groups:
- SAPIEN 3: Intermediate risk patients receiving the SAPIEN S3 valve with Commander or Certitude delivery system.
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 786
  Male | 1028
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 67
  White | 1705
  More than one race | 0
  Unknown or Not Reported | 21
Society of Thoracic Surgeons (STS) Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) Score measures patient risk of mortality or morbidity at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk of operative mortality.
  units on a scale | 4.4 (1.2)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA) functional classification of heart failure is based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
  Participants
    NYHA I | 0
    NYHA II | 682
    NYHA III | 1041
    NYHA IV | 90
    Not Assessed | 1

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Number of deaths
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- SAPIEN 3: Intermediate risk patients receiving SAPIEN S3 valve with Commander or Certitude delivery system.
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 12

2. Primary Outcome: Death
Description: Number of deaths
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 87

3. Primary Outcome: Stroke
Description: Number of participants with stroke
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 40

4. Primary Outcome: Stroke
Description: Number of participants with stroke
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 63

5. Primary Outcome: Aortic Valve Reintervention
Description: Number of participants with aortic valve reintervention
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 3

6. Primary Outcome: Aortic Valve Reintervention
Description: Number of participants with aortic valve reintervention
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 11

7. Secondary Outcome: Annular Dissection
Description: Number of participants with annular dissection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 1

8. Secondary Outcome: Aortic Dissection
Description: Number of participants with aortic dissection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 5

9. Secondary Outcome: Major Access Vascular Site Complication
Description: Number of participants with major vascular complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 20

10. Secondary Outcome: Unplanned Vascular Surgery or Intervention
Description: Number of participants with unplanned vascular surgery or intervention
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 51

11. Secondary Outcome: Retroperitoneal Bleeds
Description: Number of participants with retroperitoneal bleed
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 6

12. Secondary Outcome: Gastrointestinal Bleed
Description: Number of participants with gastrointestinal bleeding
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 2

13. Secondary Outcome: Genitourinary Bleed
Description: Number of participants with genitourinary bleeding
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 12

14. Secondary Outcome: Bleeding at Access Site
Description: Number of participants with bleeding at the access site
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | SAPIEN 3
Number analyzed (Participants) | 1814
Participants | 32

ADVERSE EVENTS:
Time Frame: All events are reported at 1 year.
Description: This trial used the TVT Registry Data Collection Form and database. On the TVT Registry Data Collection Form, clinical sites do not report the seriousness of adverse events, therefore seriousness was determined by the sponsor based on the standardized definition of a serious adverse event.
Arm/Group | SAPIEN 3
All-Cause Mortality (participants affected / at risk) | 87/1814
Serious Adverse Events (participants affected / at risk) | 818/1814
Other Adverse Events (participants affected / at risk) | 0/1814
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN 3 (N=1814)
Conduction/native pacer disturbance requiring pacemaker (Cardiac disorders) | 219 (220)
Non-valve Related Readmission (Surgical and medical procedures) | 354 (458)
Unplanned Vascular Surgery or Intervention (Surgical and medical procedures) | 53 (54)
Ischemic Stroke (Nervous system disorders) | 49 (50)
Perforation with or w/o Tamponade (Vascular disorders) | 25 (25)
Major Vascular Complication (Injury, poisoning and procedural complications) | 20 (20)
Unplanned Other Cardiac Surgery or Intervention (Surgical and medical procedures) | 29 (31)
Cardiac Arrest (Cardiac disorders) | 16 (16)
Percutaneous Coronary Intervention (Surgical and medical procedures) | 22 (22)
Myocardial Infarction (Cardiac disorders) | 17 (18)
Conduction/native pacer disturbance requiring Implantable Cardioverter Defibrillator (Cardiac disorders) | 13 (13)
Major Bleeding Event (Vascular disorders) | 32 (33)
Retroperitoneal Bleeding (Vascular disorders) | 6 (6)
Aortic Dissection (Vascular disorders) | 5 (5)
Valve Related Readmission (Surgical and medical procedures) | 15 (16)
Coronary Compression or Obstruction (Cardiac disorders) | 2 (2)
Life Threatening Bleeding (Vascular disorders) | 8 (8)
Undetermined Stroke (Nervous system disorders) | 4 (4)
New Requirement for Dialysis (Surgical and medical procedures) | 3 (3)
Hemorrhagic Stroke (Nervous system disorders) | 5 (5)
Annular Dissection (Vascular disorders) | 1 (1)
Device Embolization Left Ventricle (Vascular disorders) | 1 (1)
Aortic Valve Re-intervention (Surgical and medical procedures) | 6 (6)
Endocarditis (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-09-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT02687035/Prot_000.pdf